CLINICAL TRIAL: NCT06458816
Title: The Utility of a Non-Invasive Distractor During Arthroscopy of the Knee Joint
Brief Title: Non-Invasive Distractor During Knee Arthroscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Taylor Collaboration (Other)
Collaborators: Wilma Chan Highland Hospital Campus (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: SFORP 136
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Knee Arthritis; Knee Arthropathy
Keywords: arthroscopy; knee joint distraction; non invasive; sports medicine

STUDY DESIGN:
Intervention Model Description: This is a prospective cohort study the utility of a non-invasive distractor during arthroscopy. We hypothesize that the non-invasive distractor in conjunction with the DeMayo leg holder will provide superior medial and lateral compartment distraction with greater stability of the operative leg compared to standard manual arthroscopy techniques.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Medial Non-Invasive Knee Distraction (Experimental): medial aspect of knee with distraction device
  Interventions: Device: Non-Invasive Knee Joint Distraction
- Lateral Non-Invasive Knee Distraction (Experimental): lateral aspect of knee with distraction device
  Interventions: Device: Non-Invasive Knee Joint Distraction
- Medial Manual Knee Distraction (Active Comparator): medial aspect of knee with only manual distraction. no device.
  Interventions: Procedure: Manual Joint Distraction
- Lateral Manual Knee Distraction (Active Comparator): lateral aspect of knee with only manual distraction. no device.
  Interventions: Procedure: Manual Joint Distraction

INTERVENTIONS:
Device: Non-Invasive Knee Joint Distraction — Non-invasive Distraction device
  Arms: Lateral Non-Invasive Knee Distraction; Medial Non-Invasive Knee Distraction
Procedure: Manual Joint Distraction — no device. manual distraction.
  Arms: Lateral Manual Knee Distraction; Medial Manual Knee Distraction

SUMMARY:
Patients will be prospectively recruited for knee joint distraction who are undergoing knee arthroscopy. Patient demographics, operative factors, and rates of medical comorbidities will be collected and evaluated. Intraoperative arthroscopic images will be evaluated by the attending Orthopaedic surgeon with standard and testing mechanism and a measuring device will be used to measure the distance between the femur and tibia in the medial and lateral compartments.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age who have capacity to provide informed consent. Eligible participants will include existing patients of Dr. DiStefano who are scheduled to undergo knee arthroscopic surgery to address meniscal pathology. Study risks, benefits and description will be provided and informed consent will be obtained.

Exclusion Criteria:

* Patients with prior history of neurovascular deficiency or history of prior injury
* Patients with a prior history of knee surgery
* Patients with diagnosed knee ligament laxity or knee instability.
* Patients that are not cleared for knee arthroscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Medial Knee Joint Distraction Distance measured in millimeters (mm) during arthroscopy using a reference probe | intraoperative
  with manual distraction vs non-invasive distractor
Lateral Knee Joint Distraction Distance measured in millimeters (mm) during arthroscopy using a reference probe | intraoperative
  with manual distraction vs non-invasive distractor

SECONDARY OUTCOMES:
Pre and Post operative pain scores | preoperative and within 1 year after knee arthroscopy
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Edward De Mayo, MD, Study Director — Attending Orthopaedic Surgeon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Treuting R. Minimally invasive orthopedic surgery: arthroscopy. Ochsner J. 2000 Jul;2(3):158-63. PMID 21765685
- [Background] DeMaio M. Giants of orthopaedic surgery: Masaki Watanabe MD. Clin Orthop Relat Res. 2013 Aug;471(8):2443-8. doi: 10.1007/s11999-013-3052-1. Epub 2013 May 24. No abstract available. PMID 23703531
- [Background] Jackson RW. A history of arthroscopy. Arthroscopy. 2010 Jan;26(1):91-103. doi: 10.1016/j.arthro.2009.10.005. No abstract available. PMID 20117632
- [Background] Dienst M, Seil R, Godde S, Brang M, Becker K, Georg T, Kohn D. Effects of traction, distension, and joint position on distraction of the hip joint: an experimental study in cadavers. Arthroscopy. 2002 Oct;18(8):865-71. doi: 10.1053/jars.2002.36120. PMID 12368784
- [Background] Ohishi T, Takahashi M, Suzuki D, Matsuyama Y. Arthroscopic approach to the posterior compartment of the knee using a posterior transseptal portal. World J Orthop. 2015 Aug 18;6(7):505-12. doi: 10.5312/wjo.v6.i7.505. eCollection 2015 Aug 18. PMID 26301179
- [Background] Lee JY, Chia ZY, Jiang L, Ang B, Chang P. A Review of the Gillquist Maneuver: Modifications for a Safer and Easily Reproducible Approach for Knee Transintercondylar Notch Posterior Compartment Arthroscopy. Arthrosc Tech. 2020 Mar 3;9(4):e435-e438. doi: 10.1016/j.eats.2019.11.014. eCollection 2020 Apr. PMID 32368461
- [Background] Kramer DE, Bahk MS, Cascio BM, Cosgarea AJ. Posterior knee arthroscopy: anatomy, technique, application. J Bone Joint Surg Am. 2006 Dec;88 Suppl 4:110-21. doi: 10.2106/JBJS.F.00607. No abstract available. PMID 17142441
- [Background] Moran TE, Demers A, Awowale JT, Werner BC, Miller MD. The Outside-In, Percutaneous Release of the Medial Collateral Ligament for Knee Arthroscopy. Arthrosc Tech. 2020 Feb 25;9(3):e393-e397. doi: 10.1016/j.eats.2019.11.008. eCollection 2020 Mar. PMID 32226748
- [Background] Khademi-Kalantari K, Mahmoodi Aghdam S, Akbarzadeh Baghban A, Rezayi M, Rahimi A, Naimee S. Effects of non-surgical joint distraction in the treatment of severe knee osteoarthritis. J Bodyw Mov Ther. 2014 Oct;18(4):533-9. doi: 10.1016/j.jbmt.2013.12.001. Epub 2013 Dec 11. PMID 25440203
- [Background] Jansen MP, Mastbergen SC, van Heerwaarden RJ, Spruijt S, van Empelen MD, Kester EC, Lafeber FPJG, Custers RJH. Knee joint distraction in regular care for treatment of knee osteoarthritis: A comparison with clinical trial data. PLoS One. 2020 Jan 22;15(1):e0227975. doi: 10.1371/journal.pone.0227975. eCollection 2020. PMID 31968005
- [Background] Winkels P, Pozzi A, Cook R, Bottcher P. Prospective Evaluation of the Leipzig Stifle Distractor. Vet Surg. 2016 Jul;45(5):631-5. doi: 10.1111/vsu.12495. PMID 27357272
- [Background] Rovesti GL, Devesa-Garcia V, Urrutia PG, San Roman F, Rodriguez-Quiros J. Evaluation of a distractor to increase joint space of the stifle joint in dogs: a cadaveric study. Vet Comp Orthop Traumatol. 2015;28(3):179-85. doi: 10.3415/VCOT-14-04-0058. Epub 2015 Apr 22. PMID 25899684
- [Background] Schneider CA, Rasband WS, Eliceiri KW. NIH Image to ImageJ: 25 years of image analysis. Nat Methods. 2012 Jul;9(7):671-5. doi: 10.1038/nmeth.2089. PMID 22930834
- See also: Related Info — https://www.hilarispublisher.com/open-access/use-of-wallace-distractor-in-canine-stifle-arthroscopy-2157-7579.1000185.pdf